CLINICAL TRIAL: NCT04903184
Title: A Exploratory Phase II Clinical Trial, Double-blind, Randomized Placebo-controlled to Evaluate the Efficacy of RUTI® Against SARS-COV-2 Infection (COVID-19) in Healthcare Workers
Brief Title: Exploratory Study to Evaluate the Efficacy of RUTI® Against SARS-COV-2 Infection (COVID-19) in Healthcare Workers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: RUTI Immunotherapeutics S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RUTICOVID19-ARG
Record Dates: First submitted 2021-05-21; First posted 2021-05-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Covid-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group RUTI (Experimental): Participants will receive two dose of RUTI® vaccine at the baseline visit and after 2 weeks +/- 3 days, which will be administered subcutaneously in the deltoid region at a dose of 25 µg of fragmented, purified and liposomed heat-inactivated Mycobacterium tuberculosis bacilli in an injection volume of 0.3 mL.
  Interventions: Biological: RUTI® vaccine
- Group Placebo (Placebo Comparator): Participants will receive two dose of physiological serum will be administered subcutaneously in the deltoid region at the baseline visit and after 2 weeks +/- 3 days.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: RUTI® vaccine — Each dose of the RUTI® vaccine contains 25 µg of fragmented, purified and liposomed heat-inactivated Mycobacterium tuberculosis bacilli in a total volum of 0,3mL.
  Arms: Group RUTI
Biological: Placebo — Physiological serum, 0.9% NaCl, will be used as a placebo.
  Arms: Group Placebo

SUMMARY:
The aim of this study is to explore potential for reduction of incidence and/or morbidity of SARS-CoV-2 infection in healthcare personnel. The study will include a comparison between placebo and RUTI® vaccine in a 2:1 design.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the Informed Consent before initiating the selection procedures.
2. Population:

   1. Healthcare system workers working in contact with subjects potentially infected with SARS-CoV-2
   2. People between 18 years and 59 years
3. Willingness to meet the requirements of the protocol.
4. Negative Rapid Serological Test of SARS-CoV-2
5. The participant must agree to use effective contraceptive methods during the study period, in case of childbearing age.

Exclusion Criteria:

1. Previous SARS-CoV-2 infection
2. Pregnancy. Pregnancy test will be performed in case of doubt.
3. Breastfeeding.
4. Suspected of active viral or bacterial infection.
5. Symptoms compatible with COVID-19, despite a negative polymerase chain reaction (PCR) test.
6. Vaccination in the last 4 weeks or planned vaccination during the study period, except for influenza vaccine.
7. Participation in a research that requires experimental intervention (does not include observational studies) in the previous month before signing the Consent or during the study.
8. Severely immunocompromised people. This exclusion category includes:

   * Subjects with human immunodeficiency virus (HIV-1).
   * Neutropenic subjects with less than 500 neutrophils / mm3.
   * Subjects with solid organ transplantation.
   * Subjects with bone marrow transplantation.
   * Subjects undergoing chemotherapy.
   * Subjects with primary immunodeficiency.
   * Severe lymphopenia with less than 400 lymphocytes / mm3.
9. Malignancy, or active solid or non-solid lymphoma from the previous two years.
10. Soy allergy.
11. Direct involvement in the design or execution of the RUTICOVID19 clinical trial.
12. Retirement, transfer, long-term leave (> 1 month) due to scheduled surgery or any other event that makes it impossible to work in person at your health center during the months following the recruitment to the study.
13. Do not have a smartphone.
14. Detection by the researcher of lack of knowledge or willingness to participate and comply with all requirements of the protocol.

16. Any other findings that, at the discretion of the researcher, may compromise compliance with the protocol or that may influence significantly the interpretation or the results of the effects of the vaccine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2021-11-11 (Actual); Study Completion 2021-11-11 (Actual)

PRIMARY OUTCOMES:
Documented cumulative incidence of SARS-CoV-2 infection | 6 months
  Percent of positive serology at the end of the study or positive PCR test in the course of routine clinical practice

SECONDARY OUTCOMES:
Sick leave for SARS-CoV-2 | 6 months
  Number of days of documented sick leave for SARS-CoV-2
Days off work due to the quarantine | 6 months
  The number of days off work due to the quarantine imposed as a consequence to have acute respiratory symptoms, fever or infection documented by SARS-CoV-2
Quarantine imposed by close contact outside the center with SARS-CoV-2 positive | 6 months
  Number of days of quarantine imposed by close contact outside the center with SARS-CoV-2 positive
Fever | 6 months
  Number of days of self-reported fever (≥38 ºC)
Incidence of self-reported acute respiratory symptoms | 6 months
  Cumulative incidence of self-reported acute respiratory symptoms
Days of self-reported acute respiratory symptoms | 6 months
  Number of days of self-reported acute respiratory symptoms
Incidence of pneumonia | 6 months
  Presence of compatible symptoms and radiological or tomographic focal alteration in the context of a confirmed diagnosis of Covid-19 infection and without evidence of other concomitant pathologies
Incidence of death from SARS-CoV-2 infection | 6 months
  Cumulative incidence of death from documented SARS-CoV-2 infection
Incidence of admissions to Intensive Care Unit (ICU) | 6 months
  Cumulative incidence of admissions to intensive care unit for documented SARS-CoV-2 infection
Days in ICU | 6 months
  Number of days admitted to the ICU for documented SARS-CoV-2 infection
Incidence of mechanical ventilation | 6 months
  Cumulative incidence of need for mechanical ventilation due to documented SARS-CoV-2 infection
Incidence of hospital admissions | 6 months
  Cumulative incidence of hospital admissions for documented SARS-CoV-2 infection
Days of hospitalization | 6 months
  Number of days of hospitalization for documented SARS-CoV-2 infection
Incidence of SARS-CoV-2 antibodies | Study completion, an average of 1 year
  Incidence of SARS-CoV-2 antibodies at the end of the study period
Types of antibodies detected | Study completion, an average of 1 year
  Frequency of immunoglobulin IgG and immunoglobulin IgM
Levels of SARS-CoV-2 antibodies | Study completion, an average of 1 year
  Levels of SARS-CoV-2 antibodies

OTHER OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 6 months
  All adverse events reported by the subjects, both serious and non-serious, will be collected. All events related to a SARS-CoV-2 infection will be exempted from collection as part of the associated symptoms

CONTACTS AND LOCATIONS:
Locations (6):
- Argentina (6):
  - Hospital General de Agudos Dr. Ignacio Pirovano, Buenos Aires
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Hospital General, Mendoza
  - Hospital José Néstor Lencinas, Mendoza
  - Hospital de Clínicas Presidente Dr. Nicolás Avellaneda, San Miguel de Tucumán
  - Hospital Materno Infantil "Dr. Héctor Quintana", San Salvador de Jujuy

IPD SHARING:
Plan to Share IPD: No